CLINICAL TRIAL: NCT06567639
Title: New Insights Into Brugada Syndrome From High Density Epicardial Mapping
Brief Title: High Density Mapping in Brugada Syndrome
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Carlo de Asmundis, Prof., Universitair Ziekenhuis Brussel
Other Study IDs: BRS-EPI
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Brugada Syndrome
MeSH Terms: conditions — Brugada Syndrome | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Catheter ablation — Hybrid epicardial right ventricular (RVOT-EPI) mapping and Brugada syndrome substrate ablation technique.
  The procedure is performed in the hybrid operating room. The Advisor™ HD-Grid Mapping Catheter is delivered inside the chest through a working port and positioned under thoracoscopic view over the pulmonary artery that is consequently labeled on EAM. As a standard protocol the mapping catheter is positioned over the pulmonary artery and moved down progressively over the RVOT-EPI under continuous thoracoscopic view and at least three consecutive beats are required for each recording location point with a stable catheter position.

SUMMARY:
The current study has the following objectives:

1. To characterize the changes in amplitude and duration of epicardial right ventricular outflow tract electrograms captured through a multipolar mapping catheter in patients with Brugada syndrome before and after an ajmaline challenge.
2. To investigate the relationship between the above cited invasive electrophysiological findings and non invasive ECG imaging (ECGI) of the epicardial layer of the right ventricular outflow tract (RVOT) of patients affected by Brugada syndrome and undergoing substrate thoracoscopic catheter ablation.

DETAILED DESCRIPTION:
BACKGROUND PATHOGENESIS IN BRUGADA SYNDROME The pathophysiological basis of Brugada syndrome (BrS) is controversial. Two are the main theories which explain the electrocardiographic findings localized typically in the right precordial leads and the susceptibility of BrS patients to develop life-threatening ventricular arrhythmias: the first is that BrS is the result of a trouble in the repolarization of myocardial cells, the latter instead links BrS to depolarization and conduction abnormalities. Both theories have a common end-point in the fact that BrS patients share an anatomical and/or a functional lieu which predispose them to reentry related ventricular tachyarrhythmias and consequently to sudden cardiac death.

The repolarization theory suggests that an outward shift in the balance of currents active during phases 1 and 2 of the right ventricular (RV) epicardial action potential (AP) via either a reduction of inward current (INa or ICa) or increase in outward current (Ito, IKr, or IK-ATP) allows the intrinsically prominent Ito in RV epicardium to accentuate phase 1 repolarization. When phase 1 repolarizes to a voltage below that needed to activate the L-type Ca+2 channels, the Ca+2 channels fail to activate, resulting in loss of the AP plateau in the RV subepicardial cells where Ito is most prominent. Loss of the AP dome is commonly heterogeneous so that loss of the dome at some epicardial sites but not others creates an epicardial, as well as transmural dispersion of repolarization. Conduction of the AP dome from epicardial sites at which it is maintained to sites at which it is lost might result in the development of a closely coupled extrasystole, a phenomenon termed phase 2 reentry, which precipitates ventricular tachycardia and fibrillation (VT and VF)(1).

The depolarization hypothesis is based on the assumption that BrS patients' electrocardiographic pattern and their predisposition to develop VT/VF is related to the presence of fibrosis and to a reduced density of connexin 43 proteins in the gap-junctions of the RVOT and of other regions of the RV.

Even if both theories appear reasonable and sound, the depolarization one has obtained more consensus in the scientific community, thanks to frequent association of BrS pattern with atrioventricular conduction abnormalities and to the recent studies on epicardial mapping and radiofrequency ablation of BrS patients. The repolarization theory has been proven only in the experimental setting and is waiting for confirmation in human studies.

Two groups of scientists have shed light on the topic (i.e. epicardial mapping of BrS patient).

In their first report, Nademanee et al. showed that Brugada patients have abnormal low voltage (0.94±0.79 mV), prolonged duration (132±48 ms), and fractionated late potentials (96±47 ms beyond QRS complex) clustering in the anterior aspect of the RVOT epicardium(2). Ablation at these sites rendered VT/VF noninducible. Abnormal electrograms (EGMs) were defined as electrograms that have (1) low voltage (less than 1 mV); (2) split EGMs or fractionated EGMs with multiple potentials with at least 2 distinct components, with 20 ms isoelectric segments between peaks of individual components; and (3) wide duration (at least 80 ms) or late potentials (LPs), with distinct potentials extending beyond the end of the QRS complex. The interval from the end of the QRS complex to the end of the local electrogram was measured to determine the magnitude of LPs. Mapping and ablation were performed with NaviStar-ThermoCool catheter. A major limitation of this study was the lack of high density mapping. Second major limitation was lack of annotation to local activation (steepest negative deflection or maximum -dV/dT on unipolar) thus not allowing to distinguish between fractionation related to slow conduction or far field or other mechanisms. In order to provide an anatomical link to the above mentioned electrophysiological findings, Nademanee et al. conducted a study in post-mortem hearts of BrS patients and in parallel they provide same correlation in an in-vivo setting in patients with BrS undergoing left thoracotomy mediated radiofrequency ablation. They demonstrated that collagen is more abundant in BrS autopsied hearts compared with control hearts (odds ratio [OR]: 1.42; p = 0.026). Fibrosis was greatest in the RVOT (OR: 1.98; p = 0.003), particularly in its epicardial layer (OR: 2.00; p = 0.001). The Cx43 signal was also reduced in BrS RVOT (OR: 0.59; p = 0.001). On the other hand, in vivo RVOT samples identified epicardial and interstitial fibrosis in close anatomical association with the previously described abnormal potentials, ablation of which contributed to abolish the type 1 Brugada electrocardiogram without ventricular arrhythmia recurrence over follow-up (3). The rationale behind these anatomical findings in BrS patients is unclear: a possible explanation is that BrS is the result of an autoimmune process as shown recently by the presence of serum autoantibodies against cardiac alfa-actin, skeletal alfa-actin, keratin, and connexin-43 in a selected group of Brugada patients (4). The role of these antibodies into pathogenesis and their relationship with inflammation is yet to be extabilished (5).

The second group of scientists heavily involved in epicardial mapping of BrS patients is lead by Carlo Pappone and Joseph Brugada. In Brugada patients, they defined abnormal EGMs as those with amplitude <1.5 mV or associated wide duration (>80 ms), multiple (>3), or delayed components extending beyond the end of the QRS complex. Delay and duration of local abnormal ventricular electrograms increased after flecainide infusion in all patients. One major limitation of studies from Pappone group is the lack of high density mapping that might prevent the localization of high-frequency and low-voltage potentials (6)(7).

AIM OF THE STUDY PRIMARY OBJECTIVE To perform high density epicardial mapping of patients with Brugada syndrome before and after ajmaline injection at a standard protocol (1 mg/kg in 5 minutes) through a multipolar mapping catheter (Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ (SE) ,in association with the EnSite Precision™ Cardiac Mapping System, Abbott).

SECONDARY OBJECTIVE To evaluate the relationship between HFPs andSFPs obtained through high density invasive epicardial mapping and non invasive mapping using CardioInsightTM Noninvasive 3D Mapping System technology (Medtronic Inc, Minneapolis, MN). In brief, torso surface ECG potentials, recorded simultaneously from 250 electrodes, will be combined mathematically with patient-specific heart-torso geometry from ECG-gated computed tomography to construct epicardial potentials, unipolar EGMs, and maps of epicardial RVOT activation based on unipolar EGM LAT (9). Anatomic landmarks on computed tomographic scan will be used to define these regions: (1) left anterior descending artery separated the right ventricle (RV) and left ventricle and (2) RVOT-EPI will be defined as the region within the RV 4 cm below the pulmonary valve. Right ventricular outflow tract activation time (RVOT-AT) will be defined as the LAT of the latest RVOT-EPI point on each ECGI map.

METHODOLOGY All patients undergone high-density epicardial mapping, before and after ajmaline injection for Brugada syndrome at UZ Brussel University Hospital will be retrospectively included. In the retrospective group a multipolar mapping catheter (Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ (SE), in association with the EnSite Precision™ Cardiac Mapping System, Abbott) will be used as inclusion criteria and patients subsequently analyzed. Brugada syndrome diagnosis will be defined following current guidelines (10). All consecutive patients that will undergo to epicardial mapping and ablation for Brugada syndrome will be prospectively included. All high-density catheters (HD-grid, Abbott; PentaRay, Biosense) used in the prospective group will be included and analyzed.

Bipolar electrograms will be filtered at 30-300 Hz, noise filters on and unipolar electrograms were filtered at 0.5-100 Hz, noise filters on. For each recording location point EGM analysis will be performed from all the available dipoles within the Advisor™ HD grid, (Abbott, Minneapolis, MN) along and across splines. All EGMs will be analyzed offline using digital calipers on EnSite Precision™ Cardiac Mapping System, (Abbott, Minneapolis, MN) by two independent physicians.

STATISTICAL ANALYSIS All variables will be tested for normality with Shapiro-Wilk test. Normally distributed variables will be described as mean ± standard deviation and the groups will be compared through paired or unpaired t-test as appropriate, while the non-normally distributed variables will be described as median (Inter Quartile Range) and compared by Mann-Whitney test or Wilcoxon signed-rank test as appropriate. The categorical variables will be described as frequencies (percentages) and compared by Chi-squared test or Fisher's exact test as appropriate. Cohen's kappa test will be used to assess interobserver agreement in EGM analysis.

For all the analyses, the significance level will be set equal to 0.05. The analysis will be performed using R software version 3.6.2 (R Foundation for Statistical Computing, Vienna, Austria).

ELIGIBILITY:
Inclusion Criteria:

1. high density epicardial EAM performed with the multipolar mapping catheter Advisor™ HD-Grid Mapping Catheter, (Abbott Labs, Abbott Park, IL, USA) in association with the EnSite Precision™ Cardiac Mapping System, (Abbott Labs, Abbott Park, IL, USA);
2. epicardial EAM performed before and after ajmaline infusion at standard protocol (1 mg/kg in 5 minutes);
3. ECGI activation map performed before and after ajmaline and concomitant with invasive EAM acquisition.

Exclusion Criteria:

1. Spontaneous BrS type I pattern ECG during EAM acquisition. Patients were included if they had a history of spontaneous BrS type I;
2. other diagnosis different from BrS syndrome or overlap syndrome diagnosis by means of genetic analysis, transthoracic echocardiography, computed tomography (CT) or magnetic resonance imaging;
3. use of a different mapping catheter or mapping system;
4. history of previous BrS substrate ablation.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients who underwent hybrid thoracoscopic substrate ablation for Brugada syndrome at Universitair Ziekenhuis Brussel (UZB), between April 2018 and March 2021 will be retrospectively analyzed and included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
HD-grid electrograms | During ablation
  EGMs on HD-grid will be analyzed in detail by two physicians.

CONTACTS AND LOCATIONS:
Locations (1):
- UZB, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No